CLINICAL TRIAL: NCT03319199
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study The Effect of Combination Therapy Amino Acid L-CARNITINE and Magnesium on Fatty Liver
Brief Title: The Effect of Combination Therapy Amino Acid L-CARNITINE and Magnesium on Fatty Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawi Hazzan (Other)
Collaborators: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor-Investigator, Rawi Hazzan, Principal Investigator, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0068-16-EMC
Record Dates: First submitted 2017-10-10; First posted 2017-10-24 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary treatment Arm (Active Comparator): patients with a diagnosis of NAFDL will be randomly receive trial product "SLIM WATER" that contains L-CARNITINE and MAGNESIUM for a duration of 16 weeks.
  Interventions: Dietary Supplement: "SLIM WATER"
- Placebo Arm (Placebo Comparator): patients with a diagnosis of NAFDL will be randomly receive placebo for the initial 8 weeks and continue another 8 weeks with the trial product "SLIM WATER".
  Interventions: Other: Placebo - water

INTERVENTIONS:
Dietary Supplement: "SLIM WATER" — 2 grams of L- CARNITINE and 150 mg MAGNESIUM for a duration of 16 weeks
  Arms: Primary treatment Arm
Other: Placebo - water — for a duration of 16 weeks
  Arms: Placebo Arm

SUMMARY:
L-carnitine is an amino acid that is naturally produced in the liver and kidneys, it is involved in transporting fatty acids across the mitochondrial membrane, it could be an important component in treating a fatty liver disease.

The investigators conduct a study to evaluate the efficacy of the combination of L-Carnitine and Magnesium as a treatment for fatty liver.

DETAILED DESCRIPTION:
A phase 3, randomized, double blind placebo controlled study that evaluate the efficacy of L-Carnitine and Magnesium as a treatment for fatty liver, 60 eligible patients with a diagnosis of NAFDL will be randomly assigned in a 1:1 ratio to receive either the trial product " SLIM WATER" that contains L-CARNITINE and MAGNESIUM for a duration of 16 weeks, or placebo for the initial 8 weeks and continue another 8 weeks with the trial product "SLIM WATER". 'Follow up time is estimated to be 24 week based on monthly clinic visits and accordingly assessment of lipid profile, weight and insulin resistance.

Fibrotest will be used at the beginning of the trial and at the end (week 16) comparing the fat content before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female between the age 18 and 75.
* Patients with diagnosis of NAFLD when other etiologies for fatty liver were ruled out.
* Patients who sign a confirmed consent.

Exclusion Criteria:

* Patients with liver failure.
* Patients with acute or chronic renal failure ( CCT< 50 ml/min or creatinine > 1.5 mg/dl)
* Patients with congestive heart failure (NYHA 3-4)
* Patients with active cancer
* Patients on Estrogen therapy, MTX, chloroquine.
* Patients with a history of Hypothyroidism or Cushing disease.
* Patients who received TPN in the past 6 months.
* Patients with chronic liver disease, A1AT, Hemochromatosis, Wilson, Autoimmune, Toxic injury.
* Patients on anticoagulation therapy - Coumadin.
* Patients who use valproic acid therapy.
* Children, Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
The primary outcome is decline in serum levels of Aspartate transaminase (AST) to normal value. | 24 weeks
  Measured with blood test in IU/L
Decline in serum levels of Alanine transaminase (ALT) to normal value. | 24 weeks
  Measured with blood test in IU/L

SECONDARY OUTCOMES:
Improvement in radiological hepatic steatosis . | 24 weeks
  Liver steatosis measured by Transient Elastography - FibrsoScan done at recruitment day and at the end of treatment.
Improvement in lipid profile. | 24 weeks
  Measured with blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided